CLINICAL TRIAL: NCT00118963
Title: Effect of Repaglinide Versus Metformin Treatment in Combination With Insulin Biasp30 (Novologmix 70/30) Predinner on Glycemic and Non-Glycemic Cardiovascular Risk-Factors in Non-Obese Patients With Type-2-Diabetes With Unsatisfactory Glycaemic Control With Oral Hypoglycaemic Agents
Brief Title: Effect of Repaglinide Versus Metformin Treatment in Non-Obese Patients With Type-2-Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Steno Diabetes Center Copenhagen (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Reform
Record Dates: First submitted 2005-07-01; First posted 2005-07-12 (Estimated); Last update posted 2008-12-08 (Estimated); Status verified 2008-12

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin; repaglinide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- 3 (Active Comparator): BIAsp30 plus Metformin plus Placebo-Repaglinide. Double-Masked and randomized. Duration: 12 months.
  Interventions: Drug: Metformin; Drug: Insulin BIAsp30 (Novolog 70/30); Drug: Placebo-Repaglinide
- 2 (Active Comparator): BIAsp30 plus Repaglinide plus Placebo-Metformin. Double-masked and randomized. Duration: 12 months.
  Interventions: Drug: Insulin BIAsp30 (Novolog 70/30); Drug: Repaglinide; Drug: Placebo-Metformin
- 1 (Other): Run-in period of four months duration with Repaglinide 6 mg daily plus Metformin 2000 mg daily. No masking of interventions.
  Interventions: Drug: Metformin; Drug: Repaglinide

INTERVENTIONS:
Drug: Metformin — Tablets of 500 mg; 1000 mg two times daily.
  Arms: 1; 3
Drug: Insulin BIAsp30 (Novolog 70/30) — Subcutaneous injection. Starting dose 6 units. Titration according to glycaemic targets during the entire intervention period.
  Arms: 2; 3
Drug: Repaglinide — Tablets of 1 mg; Dosage: 2 mg three times daily.
  Arms: 1; 2
Drug: Placebo-Metformin — Tablets corresponding to 500 mg; two tablets two times daily.
  Arms: 2
Drug: Placebo-Repaglinide — Tablet corresponding to 1 mg; two tablets three times daily.
  Arms: 3

SUMMARY:
Aim:

The United Kingdom Prospective Diabetes Study (UKPDS) showed a reduction in cardiovascular events in obese patients with type-2-diabetes treated with metformin compared with other hypoglycaemic treatments with no difference in glycemic control between treatments. Non-obese patients with type-2-diabetes are usually treated with insulin-secretagogues or insulin when diet fails. Since non-obese patients with type-2-diabetes also carry a high risk of cardiovascular events, the use of metformin for this sub-group of patients might be more beneficial. Moreover, when insulin-treatment is initiated ongoing oral hypoglycaemic agents (OHA) are often continued, but in non-obese patients with type-2 diabetes little evidence exist for choosing the optimal class of OHA to be combined with insulin. The aim of the project is therefore to investigate the effect of metformin vs. an insulin-secretagogue (repaglinide) in combination with insulin on glycemic control and non-glycemic cardiovascular risk-factors in non-obese patients with type-2-diabetes, uncontrolled on diet alone.

Methodology:

Single-center, double-blind, double-dummy, randomized, parallel study involving 100 non-obese (BMI 27 kg/m2 or lower) patients with type-2-diabetes investigating the effect of treatment with metformin vs. repaglinide each in combination with biphasic insulin (Insulin-aspart 30/70, BIAsp30) for a period of 12 months.

DETAILED DESCRIPTION:
After four months run-in with repaglinide plus metformin combination-therapy, patients with HemoglobinA1c ≥6.5% will be randomized (baseline=0 month) to repaglinide 2 mg thrice-daily or metformin 1g twice-daily, both in combination with BIAsp30 (30% insulin-aspart; 70% protaminated insulin-aspart) (6U once-daily, pre-dinner) for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Non-obese patients (BMI < 27 kg/m2)
* Type 2 diabetes
* Age 40 years or older
* HbA1c = 6.5% or higher at baseline.

Exclusion Criteria:

* No known contraindications for either of the study-drugs (known allergy to the study-drugs; heart-, liver- or kidney-failure)
* Pregnancy
* Other serious physical or mental illnesses with a life-shortening prognosis.
* Drug or alcohol abuse.
* Weight-loss of more than 5 kg during the last 6 month prior to enrollment.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2003-01; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Glycemic control (HbA1c).

SECONDARY OUTCOMES:
Hypoglycaemic events
Home monitored plasma-glucose profiles
Insulin-dose
Non-glycemic cardiovascular risk factors: 24h blood-pressure measurement
24h urinary albumin excretion-rate.
Fasting and postprandial 5-point-profiles of total-cholesterol, LDL-cholesterol, HDL-cholesterol, triglycerides, free fatty acids, p-glucose, c-peptide and insulin after a standard test-meal
Markers of endothelial dysfunction, inflammation and fibrinolysis including Small-dense-LDL, Lp(a) and Apo B100, von Willebrand-factor, ICAM, VCAM, selectin, endothelin, Amadori-protein, CRP, fibrinogen, IL-6, TNF-alfa, ADMA, PAI- and t-PA-activity

CONTACTS AND LOCATIONS:
Overall Officials: Allan A Vaag, M.D. Chief Physician, Study Chair — Steno Diabetes Center Copenhagen
Locations (1):
- Steno Diabetes Center, Gentofte Municipality, Denmark

REFERENCES:
- [Derived] Lund SS, Tarnow L, Frandsen M, Nielsen BB, Hansen BV, Pedersen O, Parving HH, Vaag AA. Combining insulin with metformin or an insulin secretagogue in non-obese patients with type 2 diabetes: 12 month, randomised, double blind trial. BMJ. 2009 Nov 9;339:b4324. doi: 10.1136/bmj.b4324. PMID 19900993